CLINICAL TRIAL: NCT05709535
Title: PSMAN: POET PSMA-PET/CT Registry for High-Risk, Biochemically Relapsed, and Advanced Prostate Cancer
Brief Title: PSMA-PET/CT Registry
Status: Terminated | Type: Observational
Why Stopped: Not due to a safety concern; terminated early due to changing clinical trial landscape at centre
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: PSMA-PET-1007
Record Dates: First submitted 2023-01-19; First posted 2023-02-02 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental: [18F]PSMA-1007 Injection: A single intravenous dose of 3 - 4 MBq/kg (up to a maximum of 400 MBq) of [18F]PSMA-1007 Injection will be administered followed by PET/CT imaging.
  Interventions: Diagnostic Test: [18F]-PSMA-1007

INTERVENTIONS:
Diagnostic Test: [18F]-PSMA-1007 — [18F]PSMA-1007 is a diagnostic radiopharmaceutical for Positron Emission Tomography (PET) scan. The intervention involves single intravenous administration of [18F]PSMA-1007 for PET scan.

SUMMARY:
This is a prospective registry study to evaluate the diagnostic utility of [18F]-PSMA-1007 (PSMA-PET/CT) to stage patients with high-risk prostate cancer, localize sites of biochemical recurrence of prostate cancer, and restage patients with advanced prostate cancer before onset of new therapy.

DETAILED DESCRIPTION:
Prostate cancer is the most common non-skin malignancy and the third leading cause of cancer death in Canadian men. High-risk, recurrent, and metastatic prostate cancer is associated with poor patient outcomes. It is highly possible that the inability to accurately detect disease earlier in these patients is a key limiting factor in effectively treating patients with advanced prostate cancer.

Prostate specific membrane antigen (PSMA) is seen on many patients' prostate cancer tumours, and that PSMA expression can not only help detect cancer earlier, but it can also help determine how to treat patients with both standard treatments (e.g., surgery or radiation), as well as systemic new medical treatments (e.g. [177Lu]-PSMA-617). The new imaging technology, PSMA PET/CT, has been shown to be more sensitive and specific for the detection of metastatic prostate cancer than the current standard of care imaging (CT and bone scan) and is starting to make its way into clinical use worldwide, but is not yet available outside of clinical trials in Canada.

In recent years, prostate-specific membrane antigen (PSMA, glutamate carboxypeptidase II) has gained a resurgence of interest as a powerful imaging biomarker in prostate cancer. PSMA has been labelled with several single positron emission computed tomography (SPECT) and PET radiotracers to radiographically detect and stage the extent of disease in prostate cancer. This registry study will provide Alberta centres access to a new PET tracer, [18F]-PSMA-1007. A prospective registry study of PSMA PET/CT to guide therapy will allow enhanced access to PSMA-PET/CT and examine its effectiveness in characterizing patterns of extent, staging recurrence, and/or metastasis of high-risk prostate cancer, and to personalize therapies in men with prostate cancer. The aim is to determine the proportion of PSMA-PET/CT imaging with positive findings at local, regional, or distant sites.

ELIGIBILITY:
Inclusion Criteria:

1. Study participant has provided informed consent prior to initiation of any study specific activities/procedures.
2. Age greater than or equal to 18 years.
3. Subjects with histological diagnosis of prostate cancer.
4. Subjects with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Subjects with biochemical recurrence or persistence of prostate cancer following initial curative treatment by radical prostatectomy, with two consecutive PSA values >0.2 ng/ml measured more than 6 weeks after radical prostatectomy. If subjects received subsequent systemic therapy, the most recent PSA measurement prior to PET/CT imaging must be greater than 0.2 ng/mL OR
6. Subjects with biochemical recurrence or persistence of prostate cancer following initial curative treatment by radical prostatectomy and subsequently treated by salvage radiotherapy or pelvic node dissection, with two consecutive PSA values >0.2 ng/ml. If subjects received subsequent systemic therapy, the most recent PSA measurement prior to PET/CT imaging must be greater than 0.2 ng/mL OR
7. Subjects with biochemical recurrence of prostate cancer after initial curative therapy with radiation therapy (including brachytherapy), or non-standard local ablative therapy (such as high frequency ultrasound, cryoablation, focal laser ablation, etc.), with a PSA level >2 ng/mL above the nadir after radiation therapy OR
8. Subjects with advanced castration sensitive or castration resistant prostate cancer being considered for localized treatment (surgery, brachytherapy, radiotherapy) of recurrent or oligometastatic prostate cancer. Castration resistance is defined as a PSA level > 1.0 ng/mL, with 2 consecutive rises above the nadir, in the presence of castrate levels of testosterone (< 1.7 nmol/L) OR
9. Subjects with metastatic or castration resistant prostate cancer being evaluated for systemic therapy administered in therapeutic clinical trials. The PSA level must be > 1.0 ng/mL, with 2 consecutive rises above the nadir, in the presence of castrate levels of testosterone (< 1.7 nmol/L) OR
10. Subjects with high-risk prostate cancer, defined as T3a, Gleason ≥8, or PSA ≥20, and "very high risk" as T3b or T4 disease.
11. Patients of childbearing potential must adhere to the contraception requirement from screening throughout the study period up to 90 days after the last dose of study intervention.

Exclusion Criteria:

1. Unable to lie supine for the duration of imaging.
2. Unable to provide written consent.
3. Exceeds safe weight limit of the PET/CT bed (204.5 kg) or unable to fit through the PET/CT bore (diameter 70 cm).
4. Lack of IV access.
5. History of allergic reaction to [18F]-PSMA-1007.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: High-Risk, Biochemically Relapsed, and Advanced Prostate Cancer
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
To determine the proportion of PSMA-PET/CT imaging with positive findings at local, regional, or distant sites, utilizing a new Positron Emission Tomography (PET) tracer, [18F]-PSMA-1007 (PSMA-PET/CT). | 1 year
  The proportion of PSMA-PET/CT imaging with positive findings (whether at local, regional, or distant sites).

SECONDARY OUTCOMES:
To assess the predictive value of PSMA-PET/CT imaging on patient outcomes (e.g., radiographic/PSA progression free survival). | 1 year
  A measure such as progression-free survival in relation to subsequent oncologic treatments to assess the impact of PSMA-PET/CT imaging on patient outcomes will be calculated.
To assess the predictive value of PSMA-PET/CT imaging on patient outcomes (e.g., PSA response). | 1 year
  A measure such as best response in relation to subsequent oncologic treatments to assess the impact of PSMA-PET/CT imaging on patient outcomes will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Yip, MD, Principal Investigator — Alberta Health services
Locations (1):
- Tom Baker Cancer Centre/Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No